CLINICAL TRIAL: NCT06349694
Title: Comparison of the Efficacy of Transcutaneos Medial Plantar Nerve and Tibial Nerve Stimulation in Women With Idiopathic Overactive Bladder: A Prospective Randomized Controlled Trial
Brief Title: Comparison of the Efficacy of Transcutaneos Nerve Stimulations in Women With Idiopathic Overactive Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PamukkaleU.ftr-NYıldız-001
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Urinary Bladder, Overactive
Keywords: Idiopatic overactive bladder; Transcutaneous medial plantar nerve stimulation; Transcutaneous tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BT plus T-MPNS (Experimental): T-MPNS sessions will be performed twice a week for 6 weeks. Each session will be lasted 30 minutes. The intervention will be included a 12-session BT plus T-MPNS treatment program
  Interventions: Other: Transcutaneous MPN stimulation (T-MPNS)
- BT plus TTNS (Experimental): TTNS sessions will be performed twice a week for 6 weeks. Each session will be lasted 30 minutes. The intervention will be included a 12-session BT plus TTNS treatment program
  Interventions: Other: Transcutaneous tibial nerve stimulation (TTNS)
- BT (Control group) (Active Comparator): Information about BT will be explained to patients for 30 min. Then written form about BT will be given to be implemented as a home program.
  Interventions: Other: BT (Control group)

INTERVENTIONS:
Other: Transcutaneous MPN stimulation (T-MPNS) — Transcutaneous MPN stimulation (T-MPNS) is the electrostimulation of the lumbosacral roots that produce an activation of the lumbosacral plexus that controls the visceral organs and the pelvic floor muscles, thereby improving bladder control.
  Arms: BT plus T-MPNS
Other: Transcutaneous tibial nerve stimulation (TTNS) — Transcutaneous tibial nerve stimulation (TTNS) is the electrostimulation of the lumbosacral roots that produce an activation of the lumbosacral plexus that controls the visceral organs and the pelvic floor muscles, thereby improving bladder control.
  Arms: BT plus TTNS
Other: BT (Control group) — Conventional bladder training
  Arms: BT (Control group)

SUMMARY:
Our study is the first prospective randomized controlled trial that compares the effectiveness of transcutaneous medial plantar nerve stimulation (T-MPNS) and transcutaneous tibial nerve stimulation (TTNS) added to bladder training (BT) in women with idiopathic overactive bladder (OAB). İn this study, we aimed to assess the efficacy of T-MPNS and TTNS added to BT on quality of life (QoL) and clinical parameters asssociated with idiopathic OAB. In addition, preparation time for stimulation, treatment satisfaction and discomfort levels of the patients were evaluated.

The main questions we aim to answer are:

Is T-MPNS as effective as TTNS in the treatment of idiopathic OAB? For this purpose, we planned to compare transcutaneous applications of the tibial and plantar medial nerve in women with idiopathic OAB. 60 women with OAB will be randomized to 3 groups by using random number generator: BT program alone to Group 1 (n=20), BT plus T-MPNS to Group 2 (n=20), BT plus TTNS to Group 3 (n=20) will be applied.

DETAILED DESCRIPTION:
The main questions we aim to answer are:

Is T-MPNS as effective as TTNS in the treatment of idiopathic OAB? For this purpose, we planned to compare transcutaneous applications of the tibial and plantar medial nerve in women with idiopathic OAB. 60 women with OAB will be randomized to 3 groups by using random number generator: BT program alone to Group 1 (n=20), BT plus T-MPNS to Group 2 (n=20), BT plus TTNS to Group 3 (n=20) will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with clinical diagnosis of idiopathic OAB
* Not tolerated or unresponsive to antimuscarinics and discontinued at least 4 weeks
* Able to understand the procedures, advantages and possible side effects
* Willing and able to complate the voiding diary and QoL questionnaire
* The strength of PFM 3/5 and more

Exclusion Criteria:

* Women with stress urinary incontinence
* History of conservative therapy (BT, T-MPNS and TTNS/PTNS) within 6 months
* Pregnancy or intention to become pregnant during the study
* Current vulvovaginitis or urinary tract infections or malignancy
* Anatomic or posttraumatic malformations/skin disorders of medial plantar/tibial nerve region on inner foot/ankle that cannot allow to apply the electrodes
* More than stage 2 according to the pelvic organ prolapse quantification (POP-Q)
* Cardiac pacemaker, implanted defibrillator
* Previous urogyneceological surgery within 3 months
* Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
* Ultrasonographic evidence of PVR volume more than 100 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement in incontinence episodes (positive response rate) | Change from baseline positive response rate at the 6th week after the treatment
  Reduction in incontinence episodes will be collected from the 3-day bladder diary. Woman with ≥50% reduction in incontinence episodes were considered positive responders

SECONDARY OUTCOMES:
The severity of incontinence | Change from baseline the 24-hour pad test at the 6th week after the treatment
  The 24-hour pad test will be carried out to evaluate the severity of incontinence
Symptom severity | Change from baseline Overactive Bladder Questionnaire (OAB-V8) at the 6th week after the treatment
  Overactive Bladder Questionnaire (OAB-V8) was used to evaluate symptom severity in women with OAB
Frequency of voiding, nocturia, number of pads | Change from baseline voiding, nocturia, and the number of pads used will be collected from the 3-day bladder diary at the 6th week after the treatment
  The frequency of voiding, nocturia, and the number of pads used will be collected from the 3-day bladder diary.
Quality of life (IIQ7) | Change from baseline point of The Quality of Life-Incontinence Impact Questionnaire at the 6th week after the treatment
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7)
The Hospital Anxiety and Depression Scale (HAD) | Change from baseline point of The Hospital Anxiety and Depression Scale (HAD) at the 6th week after the treatment
  The Hospital Anxiety and Depression Scale (HAD), developed by Zigmond and Snaith in 1983, with its validity and reliability study conducted in Turkey by Aydemir et al. in 1987, assesses anxiety and depression levels. It consists of 14 questions, seven for anxiety and seven for depression, scored on a four-point Likert scale. Scores are summed for each subscale: 1, 3, 5, 7, 9, 11, and 13 for anxiety, and 2, 4, 6, 8, 10, 12, and 14 for depression. In Turkey, cutoff scores are 10/11 for anxiety and 7/8 for depression, indicating risk.
FSFI | Change from baseline point of FSFI at the 6th week after the treatment
  In the evaluation of sexual function, the FSFI questionnaire is used, consisting of 19 questions assessing six main factors: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain/discomfort. The highest possible total raw score is 95, while the lowest is 4. After multiplying the coefficients, the highest score is 36, and the lowest is 2. Impact coefficients used for scoring are: 0.6 for sexual desire, 0.3 for arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain/discomfort. An FSFI score below 26.55 is indicative of sexual dysfunction
Cure-improvement rates | Change from baseline cure and improvements at the 6th week after the treatment
  Cure and improvement rates will be recorded in all groups at the end-of-treatment assessments. Values under 1.3 g in the 24-hour pad test will be considered as "cure", while a 50% or greater reduction in wet weight compared to baseline measurements at the end of treatment will be considered as "improvement"
Treatment satisfaction | Change from baseline of their urinary incontinence on a 5-point Likert scale at the 6th week after the treatment
  The change of their urinary incontinence on a 5-point Likert scale (5, very satisfied; 1, very unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin Yıldız, Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Neurourol Urodyn. 2017 Feb;36(2):221-244. doi: 10.1002/nau.23107. Epub 2016 Dec 5. PMID 27918122
- [Background] 2. C.K. Harding, M.C. Lapitan, S. Arlandis, K. Bø, H. Cobussen-Boekhorst, E. Costantini, et al. The European Association of Urology (EAU) Guidelines. EAU Guidelines on Management of Non-Neurogenic Female Lower Urinary Tract Symptoms. In: EAU Guidelines, 2023 (Internet). Available online at: https://uroweb.org/guidelines/non-neurogenic-female-luts
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Subak LL, Quesenberry CP, Posner SF, Cattolica E, Soghikian K. The effect of behavioral therapy on urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2002 Jul;100(1):72-8. doi: 10.1016/s0029-7844(02)01993-2. PMID 12100806
- [Background] Burgio KL, Goode PS, Locher JL, Umlauf MG, Roth DL, Richter HE, Varner RE, Lloyd LK. Behavioral training with and without biofeedback in the treatment of urge incontinence in older women: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2293-9. doi: 10.1001/jama.288.18.2293. PMID 12425706
- [Background] de Groat WC, Yoshimura N. Anatomy and physiology of the lower urinary tract. Handb Clin Neurol. 2015;130:61-108. doi: 10.1016/B978-0-444-63247-0.00005-5. PMID 26003239
- [Background] de Groat WC, Griffiths D, Yoshimura N. Neural control of the lower urinary tract. Compr Physiol. 2015 Jan;5(1):327-96. doi: 10.1002/cphy.c130056. PMID 25589273
- [Background] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Background] Yildiz N, Sonmez R. Transcutaneous medial plantar nerve stimulation in women with idiopathic overactive bladder. Investig Clin Urol. 2023 Jul;64(4):395-403. doi: 10.4111/icu.20230009. PMID 37417565
- [Background] Lee HE, Cho SY, Lee S, Kim M, Oh SJ. Short-term Effects of a Systematized Bladder Training Program for Idiopathic Overactive Bladder: A Prospective Study. Int Neurourol J. 2013 Mar;17(1):11-7. doi: 10.5213/inj.2013.17.1.11. Epub 2013 Mar 31. PMID 23610706
- [Background] Schreiner L, dos Santos TG, Knorst MR, da Silva Filho IG. Randomized trial of transcutaneous tibial nerve stimulation to treat urge urinary incontinence in older women. Int Urogynecol J. 2010 Sep;21(9):1065-70. doi: 10.1007/s00192-010-1165-6. Epub 2010 May 11. PMID 20458465
- [Background] Booth J, Hagen S, McClurg D, Norton C, MacInnes C, Collins B, Donaldson C, Tolson D. A feasibility study of transcutaneous posterior tibial nerve stimulation for bladder and bowel dysfunction in elderly adults in residential care. J Am Med Dir Assoc. 2013 Apr;14(4):270-4. doi: 10.1016/j.jamda.2012.10.021. Epub 2012 Nov 30. PMID 23206722
- [Background] Tezer T, Yildiz N, Sarsan A, Alkan H. Short-term effect of magnetic stimulation added to bladder training in women with idiopathic overactive bladder: A prospective randomized controlled trial. Neurourol Urodyn. 2022 Aug;41(6):1380-1389. doi: 10.1002/nau.24957. Epub 2022 May 20. PMID 35593007
- [Background] Yamanishi T, Homma Y, Nishizawa O, Yasuda K, Yokoyama O; SMN-X Study Group. Multicenter, randomized, sham-controlled study on the efficacy of magnetic stimulation for women with urgency urinary incontinence. Int J Urol. 2014 Apr;21(4):395-400. doi: 10.1111/iju.12289. Epub 2013 Oct 14. PMID 24118165
- [Background] Firinci S, Yildiz N, Alkan H, Aybek Z. Which combination is most effective in women with idiopathic overactive bladder, including bladder training, biofeedback, and electrical stimulation? A prospective randomized controlled trial. Neurourol Urodyn. 2020 Nov;39(8):2498-2508. doi: 10.1002/nau.24522. Epub 2020 Sep 22. PMID 32960999
- [Background] O'Sullivan R, Karantanis E, Stevermuer TL, Allen W, Moore KH. Definition of mild, moderate and severe incontinence on the 24-hour pad test. BJOG. 2004 Aug;111(8):859-62. doi: 10.1111/j.1471-0528.2004.00211.x. PMID 15270937
- [Background] 19. Tarcan T, Mangır N, Özgür MÖ, Akbal C. OAB-V8 Overactive Bladder Questionnaire Validation Study. (Turkish) Üroloji Bülteni 2012;21:113-116. http://www.kontinansdernegi.org/userfiles/media/kontinans.galenos.com.tr/oab-v8-asiri-aktif-mesane-sorgulama-formu.pdf
- [Background] Acquadro C, Kopp Z, Coyne KS, Corcos J, Tubaro A, Choo MS, Oh SJ. Translating overactive bladder questionnaires in 14 languages. Urology. 2006 Mar;67(3):536-40. doi: 10.1016/j.urology.2005.09.035. PMID 16527574
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117